CLINICAL TRIAL: NCT02942251
Title: The Study of Relapse Predicting Model for First Episode Depression: Big Data Analysis Based on Clinical Features and Immunochemistry
Brief Title: Relapse Predicting Model for First Episode Depression
Acronym: RPM-FED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pending
Record Dates: First submitted 2016-10-20; First posted 2016-10-24 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Major Depressive Disorders
Keywords: MDD; big data analytics
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Dosage Forms; Transplantation Immunology; Comorbidity; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Clinical features and medication (Experimental): A group patients with significant high risk of clinical features and medications.
  Interventions: Other: Clinical features and medication
- Psycho-social (Experimental): A group patients with significant high risk of psycho-social problems.
  Interventions: Other: Psycho-social
- immunology (Experimental): A group patients with significant high risk of immune disturbance.
  Interventions: Other: immunology
- Laboratory abnormality (Experimental): A group patients with significant high risk of Laboratory abnormalities.
  Interventions: Other: Laboratory abnormality
- Comorbidity (Experimental): A group patients with physical or mental disorders comorbidities.
  Interventions: Other: Comorbidity
- Treatment as usual (Experimental): Control group.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: Clinical features and medication — This group will be suggested to take optimize treatment according to Chinese treatment guidelines.
  Arms: Clinical features and medication
Other: Psycho-social — This group will be suggested to add on psychotherapy on medical treatment.
  Arms: Psycho-social
Other: immunology — This group will be suggested to add on Omega-3 polyunsaturated fatty acid(PUFAs) on medical treatment.
  Arms: immunology
Other: Laboratory abnormality — This group will be suggested to more safety antidepressants.
  Arms: Laboratory abnormality
Other: Comorbidity — This group will be suggested to treat their comorbidities as well as treat MDD.
  Arms: Comorbidity
Other: Treatment as usual — Patients will accept routine treatments based on psychiatrist experience, not based on the relapse predict model.
  Other Names: Treatment as usual(TAU)
  Arms: Treatment as usual

SUMMARY:
Major depressive depression(MDD) is an severe public mental disorders. The purpose of current study is using big data analysis based on clinical features and immunochemistry to investigate and establish an relapse predict model for patients with first episode MDD.

DETAILED DESCRIPTION:
Major depressive depression(MDD) is an severe public mental disorders. The purpose of current study is using big data analysis based on clinical features and immunochemistry to investigate and establish an relapse predict model for patients with first episode MDD.

This study includes two steps. Step 1: Big data analysis based on the clinical features and immunochemical figures of 30000 patients with first episode MDD will be conducted to construct a relapse predict model.

Step 2: 300 patients with first episode MDD will be recruited in this step. Physicians prefer to give corresponding treatment recommendation based on the predictive factors to verify this relapse model.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years old;
* Han Chinese;
* Outpatient and inpatient patients;
* Patients met Diagnostic and Statistical Manual of Mental Disorders(DSM-IV-TR) criteria of bipolar I or II disorder, currently depressed, ascertained with the Mini International Neuropsychiatric Interview (MINI)
* Hamilton Depression Scale(HAM-D) total score≥17, HAM-D item 1 (depressed mood) score≥2, and Young Mania Rating Scale(YMRS) total score≤10 at baseline;
* Written informed consent was given;
* Junior high school education and above, with enough audio-visual ability to accomplish the visits;
* Normally resident in one country and had a residential address, able to follow-up.

Exclusion Criteria:

* Bipolar disorder rapid cycling or mixed episode;
* Experienced DSM-IV-TR axis I disorders in the 6 months prior to randomization;
* Severe personality disorder, metal retardation, anorexia/bulimia nervosa;
* Actively suicide ascertained by research psychiatrist or HAM-D item 3 score≥3(suicidality);
* Female patients who were pregnant, planning to be pregnant or breast feeding;
* Severe medical or neurological problems.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
HAM-D total score | 12 weeks
  The change from baseline to end of study (EOS) in HAM-D total score

SECONDARY OUTCOMES:
Time to relapse | 12 months
  The time to new intervention for an emerging mood episode

CONTACTS AND LOCATIONS:
Overall Officials: Jun Chen, M.D., Ph.D, Principal Investigator — Shanghai Mental Health Center

IPD SHARING:
Plan to Share IPD: Undecided